CLINICAL TRIAL: NCT05163496
Title: A Randomized, Placebo-controlled Trial of Psychedelic-assisted Psychotherapy With Single Dose Psilocybin for Frontline Clinicians Experiencing COVID-related Symptoms of Depression and Burnout
Brief Title: Frontline Clinician Psilocybin Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Anthony Back MD, Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00013891
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Burnout, Caregiver; Burnout, Professional; COVID-19; Depression; Post Traumatic Stress Disorder; Moral Injury
Keywords: psilocybin; psychedelic assisted psychotherapy
MeSH Terms: conditions — Caregiver Burden; Burnout, Professional; COVID-19; Depression; Stress Disorders, Post-Traumatic | interventions — Psilocybin

STUDY DESIGN:
Intervention Model Description: This study tests a hypothesis that a single session of psilocybin (the 'medication dosing' session) in the context of pre- and post-dose psychotherapy will result in improvement of symptoms of depression and burnout measured 4 weeks post-dose. This study hypothesis will be tested in a single site, double-blind, randomized controlled design involving 30 clinician participants that will compare effects of a single 25mg oral dose of psilocybin to a 250 mg of niacin (active placebo). The primary outcome measurements will be collected 4 weeks after the psilocybin dose, after which the participant group assignment will be unblinded, and participants who received niacin will be offered the opportunity to have a second dose session with a 25 mg dose (with pre- and post-dose psychotherapy).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The investigators, study therapists, and outcomes assessors will all be blinded in the randomized phase of the study. Participants will be unblinded after the primary outcome, and those receiving placebo will be eligible to receive open label psilocybin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psilocybin arm (Experimental): psychedelic assisted psychotherapy + 25mg psilocybin
  Interventions: Drug: Psilocybin (Usona Institute)
- Placebo (Active Comparator): Psychedelic assisted psychotherapy + 250mg niacin
  Interventions: Drug: Active placebo

INTERVENTIONS:
Drug: Psilocybin (Usona Institute) — PAP + psilocybin 25 mg
  Other Names: Psychedelic-assisted psychotherapy (PAP)
  Arms: Psilocybin arm
Drug: Active placebo — PAP + niacin 250mg
  Other Names: PAP with placebo
  Arms: Placebo

SUMMARY:
This study aims to investigate the effects of a single dose of psilocybin, delivered in the contextof pre- and post-dose psychotherapy, on symptoms of depression and burnout suffered by healthcare clinicians as a result of frontline work in the COVID pandemic.

DETAILED DESCRIPTION:
Aim 1:

To assess short- and longer-term effects of psilocybin-assisted psychotherapy (PAP) on symptoms of depression experienced by physicians and nurses with frontline work exposure in the COVID pandemic.

Hypothesis 1.1: Compared to active placebo, PAP will result in short term improvement in symptoms of depression 1 day and 1 week after the psilocybin dose session. Hypothesis 1.2: Compared to active placebo, PAP will result in longer term improvement of symptoms of depression 4 weeks after the medication dosing session. The primary outcome will be a comparison between the psilocybin 25 mg vs control groups of a combination of depression symptoms measured at 4 weeks post medication dose session. 1.1.2. Aim 2: To explore short- and longer-term effects of psilocybin-assisted psychotherapy (PAP) on symptoms of burnout experienced by physicians and nurses with frontline work exposure in the COVID pandemic. Hypothesis 2.1: Compared to active placebo, PAP will result in short term improvement in symptoms of burnout 1 day and 1 week after the psilocybin dose session.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be physicians or nurses with at least 1 month of frontline clinical experience during the COVID pandemic who rate at least 2 of 4 items from the COVID Exposure index as 'more than half the days' during their peak 2 week period of exposure: i. Caring for someone critically ill with COVID-19, or who became critically ill while you were involved; ii. Working longer hours than usual in order to provide assistance or care to individuals with COVID-19; iii. Witnessing or responding to a death related to COVID-19, or losing a patient you had been caring for to COVID-19; iv. Caring for patients who have died without family physically present due to COVID-19 precautions
2. Have a Montgomery-Asberg Depression Rating Scale (MADRS) clinician-administered depression score >21, indicating moderately severe symptoms.
3. Have had persistent symptoms despite at least one medication and/or therapy trial of standard care treatment for depression.
4. English speaking - able to understand the process of consent and the risk and benefits associated with the study, and able to give written informed consent.
5. Must be willing to sign a medical release for the investigators to communicate directly with their therapist and doctors to confirm a medication and/or medical history. This is decided on a case-by-case basis upon the discretion of the PI.
6. Must be driven home after the medication dosing session by a driver (which could be a friend, family, rideshare or taxi).
7. Must provide at least one adult to have continuous contact with the participant, provide participant transportation, monitor changes in the participant's behavior, and notify research staff of behavior changes.
8. Has been off selective serotonin inhibitors (SSRIs) for at least five half-lives of the drug plus 2 weeks.
9. Must avoid taking any psychiatric medications or starting a new psychiatric medication during the study. Should participant's doctor recommend starting a new psychiatric medication, participant will be required to notify the study team and the subject would withdraw from the study
10. Must provide a contact (relative, spouse, close friend or other caregiver) who is willing and able to be reached by the Clinical Investigators in the event of a participant becoming suicidal.
11. If able to bear children, must have a negative pregnancy test at study entry.
12. Are willing to commit to preparation sessions, medication dosing sessions, integration sessions, to complete evaluation instruments and commit to be contacted for all necessary telephone contacts.

Exclusion Criteria:

1. Personal or immediate family history of schizophrenia, bipolar affective disorder, delusion disorder, paranoid disorder, or schizoaffective disorder.
2. Suicidal ideation with a Columbia Suicide Severity Rating Scale (C-SSRS) > 3
3. Current substance abuse disorder (except in the case of mild alcohol use )
4. Neuroleptic and SSRI medications that cannot be tapered and discontinued in conjunction with the participant's prescribing physician.
5. Unstable neurological or medical condition; history of seizure, chronic/severe headaches.
6. Positive urine pregnancy test at the time of screening
7. Any unstable medical condition that my render study procedures unsafe.
8. Any use of psychedelic drugs within the prior 12 months.
9. Use of tramadol, due to the potential for serotonin syndrome with concomitant use of psilocybin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2024-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Back, MD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: We anticipate sharing these data starting with publication of study results and for at least 3 years.
Access Criteria: To be determined.

REFERENCES:
- [Derived] Back AL, Freeman-Young TK, Morgan L, Sethi T, Baker KK, Myers S, McGregor BA, Harvey K, Tai M, Kollefrath A, Thomas BJ, Sorta D, Kaelen M, Kelmendi B, Gooley TA. Psilocybin Therapy for Clinicians With Symptoms of Depression From Frontline Care During the COVID-19 Pandemic: A Randomized Clinical Trial. JAMA Netw Open. 2024 Dec 2;7(12):e2449026. doi: 10.1001/jamanetworkopen.2024.49026. PMID 39636638

RESULTS

PARTICIPANT FLOW:
Groups:
- Psilocybin Arm; Open-label Psilocybin (for Placebo Participants): 2 preparation therapy sessions, then a medication session with 25mg psilocybin, then 3 integration therapy sessions. The psilocybin was provided by the Usona Institute.
- Placebo: 2 preparation therapy sessions, then a medication session with niacin 100 mg, then 3 integration therapy sessions. The niacin was provided by the Usona Institute.
Period: Randomized Phase
Arm/Group | Psilocybin Arm | Placebo | Open-label Psilocybin (for Placebo Participants)
Started | 15 | 15 | 0
Completed | 15 | 15 | 0
Not Completed | 0 | 0 | 0
Period: Open Label Phase
Arm/Group | Psilocybin Arm | Placebo | Open-label Psilocybin (for Placebo Participants)
Started | 0 | 0 | 12
Completed | 0 | 0 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: To be eligible, clinicians had to have more than 1 month of direct frontline clinical care experience and had to endorse at least 2 of 4 items from a COVID-19 occupational exposure index as occurring more than half of the day during that time.
Groups:
- Total: Total of all reporting groups
Arm/Group | Psilocybin Arm | Placebo | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 15 | 15 | 30
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 40 [29 to 60] | 36 [30 to 48] | 38 [29 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 7 | 8 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Montgomery-Asberg Depression Rating Scale
Description: Assesses symptoms of depression (clinician-assessed): minimum score 0, max 60; higher score indicates more severe symptoms
Time Frame: 4-weeks post psilocybin-assisted psychotherapy
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Psilocybin Arm | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | 21.33 (7.84) | 9.33 (7.32)
Statistical Analysis 1: Comparison: Psilocybin Arm vs Placebo; The null hypothesis was that the mean change in MADRS score from the preparation 1 session to day 28 would be the same in both niacin and psilocybin groups. The alternative hypothesis was that the change in the psilocybin group would be greater than the change in the niacin group, with an assumed true effect size of 1.06 SD units based on findings in prior studies. With 15 participants per group, this study had 80% power to observe a statistically significant difference between groups; Test type: Superiority; p < .001, t-test, 2 sided; Mean Difference (Net) = 12.00, Standard Deviation .80

2. Secondary Outcome: Montgomery-Asberg Depression Rating Scale
Description: as for outcome 1
Time Frame: 24 weeks post-psilocybin in the randomized phase psilocybin arm
Population: Participants in the placebo arm were not followed with the MADRS score after Day 28
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psilocybin Arm | Placebo
Number analyzed (Participants) | 15 | 0
score on a scale | 3.67 (4.48) |

3. Secondary Outcome: Stanford Fulfillment Index
Description: Assesses professional burnout in 3 components that are scored separately (professional fulfillment, interpersonal disengagement, work exhaustion)
Time Frame: 1,4,8,12,24 -weeks post psilocybin-assisted psychotherapy
Reporting Status: Not Posted

4. Secondary Outcome: PTSD Checklist for DSM-5 (PCL5)
Description: Assesses symptoms of post-traumatic stress disorder; minimum score 0, max 80; higher scores indicate more severe symptoms of PTSD
Time Frame: 4 weeks post-psilocybin or placebo session
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Psilocybin Arm | Placebo
Number analyzed (Participants) | 15 | 15
score on a scale | 16.67 (15.04) | 6.74 (10.69)

5. Secondary Outcome: Moral Injury Symptom Scale
Description: Assesses symptoms of moral injury: minimum score 10, max 100; higher score indicates more severe symptoms
Time Frame: 4, 24 weeks post-psilocybin-assisted psychotherapy
Reporting Status: Not Posted

6. Secondary Outcome: Beck Depression Index
Description: Assess self-reported symptoms of depression: minimum score 0, max 63; higher score indicates more severe symptoms of depression
Time Frame: 1, 4, 8, 12, 24-weeks post-psilocybin-assisted psychotherapy
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months after intervention was completed
Description: Definitions are the same as clinicaltrials.gov
Groups:
- Open-label Psilocybin (for Placebo Participants): psychedelic assisted psychotherapy + 25mg psilocybin
  Psilocybin (Usona Institute): PAP + psilocybin 25 mg
Arm/Group | Psilocybin Arm | Placebo | Open-label Psilocybin (for Placebo Participants)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/12
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT05163496/Prot_SAP_000.pdf